CLINICAL TRIAL: NCT07074678
Title: Prognostication of Recovery in Early Disorders of Consciousness Study
Acronym: PREDICT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, David Fischer, Principal Investigator, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 852381; 1K23NS136745-01A1 (NIH)
Record Dates: First submitted 2025-05-22; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Disorder of Consciousness; Comatose; Coma; Prolonged; Vegetative State; Minimally Conscious State
MeSH Terms: conditions — Consciousness Disorders; Coma; Persistent Vegetative State | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Patients and healthy controls will undergo functional MRI, which may include auditory and noxious stimulation.
  Interventions: Diagnostic Test: Functional MRI (fMRI)

INTERVENTIONS:
Diagnostic Test: Functional MRI (fMRI) — Research MRI, which will include both structural and functional sequences, will either be collected independently, or in conjunction with clinically-indicated sequences. Functional MRI captures the blood oxygen level dependent (BOLD) signal that reflects brain activity. A subset of the PREDICT study fMRI will include sequences with auditory and/or noxious stimulation. Noxious stimulation will be delivered with an MRI-compatible device that delivers intermittent nailbed pressure under computerized control. Additionally, the BOLD signal will be captured at rest to investigate functional neural networks.

SUMMARY:
The goal of this study is to determine the extent to which neuroimaging metrics (e.g., functional MRI) are associated with the current level of consciousness, and future consciousness recovery, in patients with disorders of consciousness resulting from acute brain injury. The main questions this study aims to answer are:

How do functional MRI findings (e.g., covert consciousness and network connectivity) associate with current level of consciousness? How do functional MRI findings (e.g., covert consciousness and network connectivity) associate with future recovery of consciousness? How does noxious stimulation affect the detection of covert consciousness and functional brain network connectivity?

DETAILED DESCRIPTION:
Patients with disorders of consciousness (lacking overt signs of consciousness such as command-following) due to acute brain injury will be identified and enrolled via the Recovery of Consciousness Via Evidence-Based Medicine and Research (RECOVER) Program. Patients in the study will undergo a detailed behavioral consciousness assessment (with the Coma Recovery Scale - Revised [CRS-R]), conducted by specially trained personnel, as well as a task-based functional MRI with auditory stimulation (motor commands) to assess for technologic covert consciousness (the willful modulation of brain activity to command) and functional brain network connectivity. For a subset of patients, the functional MRI will be performed with and without noxious stimulation, during the same scanning session. Patients will undergo repeat behavioral evaluations at hospital discharge, and 3 and 6 months after, to assess for overt consciousness recovery.

ELIGIBILITY:
For patients:

Inclusion Criteria:

* Acute brain injury (including, but not limited to ischemic stroke, intracranial hemorrhage, anoxic brain injury, traumatic brain injury, or encephalitis)
* Inability to follow commands due to a disorder of consciousness (comatose, vegetative, or minimally conscious state) caused by the underlying brain injury
* Age 18 or greater
* Enrolled within 28 days of brain injury

Exclusion Criteria:

* Imminent death (as indicated, for example, by planned transition to palliative measures, brain death testing, or severe medical instability)
* MRI contraindications would exclude patients from imaging component of study

For healthy controls:

Exclusion Criteria:

* MRI contraindications
* History of brain injury to neurological disease
* History of diabetes, high blood pressure, kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2028-03-08 (Estimated); Study Completion 2029-03-08 (Estimated)

PRIMARY OUTCOMES:
Detection of technologic covert consciousness | Baseline, during hospitalization (estimated approximately 1 month from brain injury)
  Brain activity during the delivery of commands, as compared to brain activity during rest, will be measured during the functional MRI scan. Brain activity that is significantly more associated with commands and that occurs in the premotor cortex or supplementary motor area will be interpreted as evidence of technologic covert consciousness.
Functional network connectivity | Baseline, during hospitalization (estimated approximately 1 month from brain injury)
  Functional connectivity of brain networks will be measured during a resting state functional MRI sequence without noxious stimulation. Another sequence may be obtained during noxious stimulation.
Detection of behavioral covert consciousness | Baseline, during hospitalization (estimated approximately 1 month from brain injury), within 24 hours of the functional MRI
  The Coma Recovery Scale - Revised (CRS-R) will be used to assess the presence of behavioral covert consciousness, defined as the minimally conscious state minus (non-language based, but purposeful, behaviors), or the minimally conscious state plus (command-following, intelligible verbalization, and intentional communication). Higher scores (maximum 23) reflect higher levels of consciousness than lower scores (minimum 0).
Overt consciousness recovery based on Disability Rating Scale | Through study completion: At hospital discharge (estimated approximately 1 month from brain injury), 3 months after hospital discharge, and 6 months after hospital discharge
  Overt consciousness, defined as command-following as measured with the Disability Rating Scale, will be evaluated at hospital discharge, and 3 and 6 months afterwards.

CONTACTS AND LOCATIONS:
Overall Officials: David J Fischer, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided